CLINICAL TRIAL: NCT04543955
Title: Study of Telotristat (Xermelo) in Combination With Luetetium Lu177 Dotatate (Lutathera) in Well-Differentiated Neuroendocrine Tumors
Brief Title: Telotristat With Lutathera in Neuroendocrine Tumors
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor cancelled research
Sponsor: Lowell Anthony, MD (Other)
Collaborators: TerSera Therapeutics LLC (Industry)
Responsible Party: Sponsor-Investigator, Lowell Anthony, MD, Professor, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MCC-20-GI-114-PMC
Record Dates: First submitted 2020-09-02; First posted 2020-09-10 (Actual); Results first posted 2023-06-27 (Actual); Last update posted 2023-06-27 (Actual); Status verified 2023-06

CONDITIONS: Neuroendocrine Tumors
Keywords: NET
MeSH Terms: conditions — Neuroendocrine Tumors | interventions — telotristat; telotristat ethyl

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm 1: Low-Dose Telotristat (Experimental): Participants in this group will receive 750mg Telotristat per day.
  Interventions: Drug: Telotristat (Low-Dose)
- Arm 2: High-Dose Telotristat (Experimental): Participants in this group will receive 1500mg Telotristat per day.
  Interventions: Drug: Telotristat (High-Dose)

INTERVENTIONS:
Drug: Telotristat (Low-Dose) — Participants in this group will receive Lutetium Lu 177 Dotate (Lutathera) by IV every 2 months (Q8weeks) for a total of 4 doses. They will also receive oral Telotristat at 750mg per day (250mg TID) for 20 months.
  Other Names: Xermelo
  Arms: Arm 1: Low-Dose Telotristat
Drug: Telotristat (High-Dose) — Participants in this group will receive Lutetium Lu 177 Dotate (Lutathera) by IV every 2 months (Q8weeks) for a total of 4 doses. They will also receive oral Telotristat at 1500mg per day (500mg TID) for 20 months.
  Other Names: Xermelo
  Arms: Arm 2: High-Dose Telotristat

SUMMARY:
This trial will test the hypothesis that Telotristat treatment increases the antitumor efficacy of Lutetium Lu 177 Dotatate therapy in neuroendocrine tumors (NETs).

DETAILED DESCRIPTION:
Neuroendocrine tumors (NETs) are a very heterogeneous group of tumors that develop predominantly in the gastrointestinal and pulmonary systems. Clinical detection and diagnosis are more reliable at late stages when metastatic spread has occurred. Patients with advanced disease may suffer from complications of uncontrolled hormone secretion and usually succumb due to tumor progression.

This trial tests the hypothesis that inhibition of serotonin production with Telotristat will lead to cytostatic effects on neuroendocrine tumors and will complement the anti-tumor activity of Lutetium 177 Dotatate. The proposed combination may result in improved treatment efficacy as reflected by improved 20-month progression-free survival (PFS) as compared to historical control.

ELIGIBILITY:
Inclusion Criteria:

* Metastatic, or unresectable, histologically confirmed well-differentiated grade 1 and 2 neuroendocrine tumor with a positive gallium 68 Dotatate scan within 6 months prior to study enrollment
* Baseline CT scan or MRI with measurable progressive disease based on RECIST Criteria
* Failure of at least one prior systemic cancer treatment for this diagnosis
* Recovered from Adverse Events of previously administered therapeutic agents to Grade 2 or less toxicity according to CTCAE version 5.0
* Eastern Cooperative Oncology Group (ECOG) performance status ≤2
* normal organ and marrow function

Exclusion Criteria:

* Prior exposure to Lutetium Lu 177 Dotatate
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to Telotristat or Lutetium Lu 177 Dotatate.
* Presence of unstable angina or myocardial infarction
* New York Heart Association (NYHA) Class III or IV heart failure
* uncontrolled angina
* history of severe coronary artery disease, severe uncontrolled ventricular arrhythmias, sick sinus syndrome, or electrocardiographic evidence of acute ischemia or Grade 3 conduction system abnormalities
* Pregnant or lactating women
* Women of childbearing potential or male patients of reproductive potential
* Any other significant medical or psychiatric condition, currently uncontrolled by treatment, which may interfere with completion of the study

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2021-09-13 (Actual); Primary Completion 2022-06-03 (Actual); Study Completion 2022-06-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lowell Anthony, MD, Principal Investigator — University of Kentucky
Locations (1):
- Markey Cancer Center, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm 1: Low-Dose Telotristat | Arm 2: High-Dose Telotristat
Started | 1 | 0
Completed | 0 | 0
Not Completed | 1 | 0
Not completed — Company cancelled study | 1 | 0

BASELINE CHARACTERISTICS:
Population: Research cancelled and 0 participants enrolled in Arm 2
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1: Low-Dose Telotristat | Arm 2: High-Dose Telotristat | Total
Number analyzed (Participants) | 1 | 0 | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 |  | 0
  Between 18 and 65 years | 0 |  | 0
  >=65 years | 1 |  | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 |  | 1
  Male | 0 |  | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 |  | 0
  Asian | 0 |  | 0
  Native Hawaiian or Other Pacific Islander | 0 |  | 0
  Black or African American | 0 |  | 0
  White | 1 |  | 1
  More than one race | 0 |  | 0
  Unknown or Not Reported | 0 |  | 0
Region of Enrollment [Number; unit: participants]
  United States | 1 |  | 1

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival (PFS)
Description: Progression-free survival at 20 months.
Time Frame: 20 months
Population: One participant was enrolled in this study. Due to the possibility that participants could reasonably be identified due to low enrollment, data cannot be presented.
Arm/Group | Arm 1: Low-Dose Telotristat | Arm 2: High-Dose Telotristat
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Overall Response Rate (ORR)
Description: Overall response rate using RECIST v1.1 at 6 and 12 months after therapy
Time Frame: 6 and 12 months
Population: as for outcome 1
Arm/Group | Arm 1: Low-Dose Telotristat | Arm 2: High-Dose Telotristat
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Median Progression-Free Survival (PFS)
Description: Median progression-free survival.
Time Frame: 36 month
Population: as for outcome 1
Arm/Group | Arm 1: Low-Dose Telotristat | Arm 2: High-Dose Telotristat
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Urinary 5-HIAA
Description: Levels of urinary 5-Hydroxyindoleacetic acid (5-HIAA) will be measured at baseline and 12 months.
Time Frame: Baseline and 12 months
Population: as for outcome 1
Arm/Group | Arm 1: Low-Dose Telotristat | Arm 2: High-Dose Telotristat
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Quality of Life (QLQ-C30)
Description: The Quality of Life Questionnaire C30 (QLQ-C30) was developed by the European Organization for Research and Treatment of Cancer (EORTC) to assess quality of life in cancer patients.It includes five function domains (physical, emotional, social, role, cognitive), eight symptoms (fatigue, pain, nausea/vomiting, constipation, diarrhea, insomnia, dyspnea, and appetite loss), as well as global health/quality-of-life and financial impact. Subjects respond on a four-point scale from "not at all" to "very much" for most items.Raw scores are linearly converted to a 0-100 scale with higher scores reflecting higher levels of function and higher levels of symptom burden.
Time Frame: 20 month
Population: as for outcome 1
Arm/Group | Arm 1: Low-Dose Telotristat | Arm 2: High-Dose Telotristat
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Quality of Life (QLQ-GI.NET21)
Description: The Quality of Life GI Neuroendocrine Tumor survey (QLQ-GINET21) contains a total of 21 items: four single-item assessments relating to muscle and/or bone pain (MBP), body image (BI), information (INF) and sexual functioning (SX), together with 17 items organised into five proposed scales: endocrine symptoms (ED; three items), GI symptoms (GI; five items), treatment-related symptoms (TR; three items), social functioning (SF) and disease-related worries (DRW; three items). The response format of the questionnaire is a four-point Likert scale. Responses are linearly transformed to a 0-100 scale using EORTC guidelines, with higher scores reflecting more severe symptoms.
Time Frame: 20 month
Population: as for outcome 1
Arm/Group | Arm 1: Low-Dose Telotristat | Arm 2: High-Dose Telotristat
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Only 1 participant was enrolled in this study. Based on the low enrolment number, no data is reported here in order to protect and maintain participant privacy/confidentiality.
Description: Only 1 participant was enrolled in this study. Based on the low enrolment number, no data is reported here in order to protect and maintain participant privacy/confidentiality.
Arm/Group | Arm 1: Low-Dose Telotristat | Arm 2: High-Dose Telotristat
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-04-11): https://cdn.clinicaltrials.gov/large-docs/55/NCT04543955/Prot_SAP_000.pdf